CLINICAL TRIAL: NCT03950076
Title: EdoxabaN for IntraCranial Hemorrhage Survivors with Atrial Fibrillation (ENRICH-AF)
Acronym: ENRICH-AF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENRICH-AF
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Hemorrhages; Atrial Fibrillation
Keywords: Edoxaban; Intracranial Hemorrhage; Hemorrhagic Stroke
MeSH Terms: conditions — Intracranial Hemorrhages; Atrial Fibrillation; Hemorrhagic Stroke | interventions — edoxaban

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open, blinded end-point (PROBE), multicenter international trial
Who Masked: Outcomes Assessor
Masking Description: open label study where outcomes assessor is blinded to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Edoxaban 60/30mg daily (Experimental): Edoxaban 60/30 mg daily (lower dose depending on clinical criteria)
  Interventions: Drug: Edoxaban
- Non-anticoagulant medical therapy (Active Comparator): Non-anticoagulant medical therapy: no antithrombotic therapy or antiplatelet monotherapy (at discretion of local investigator)
  Interventions: Other: Non-anticoagulant medical therapy

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 60mg (or 30mg as determined by clinical criteria)
  Other Names: Lixiana; Savaysa
  Arms: Edoxaban 60/30mg daily
Other: Non-anticoagulant medical therapy — Non-anticoagulant medical therapy as determined by the local investigator includes i) No antithrombotic therapy ii) Antiplatelet monotherapy, including de novo indication for antiplatelet monotherapy during course of the study
  Arms: Non-anticoagulant medical therapy

SUMMARY:
To assess whether edoxaban (60/30 mg daily) compared to non-antithrombotic medical therapy (either no antithrombotic therapy or antiplatelet monotherapy) reduces the risk of stroke (composite of ischemic, hemorrhagic and unspecified stroke) or systemic embolism in high-risk atrial fibrillation (CHA2DS2-VASc ≥2) patients with previous intracranial hemorrhage.

DETAILED DESCRIPTION:
The EdoxabaN foR IntraCranial Hemorrhage survivors with Atrial Fibrillation (ENRICH-AF) study is a prospective, randomized open-label, blinded end-point (PROBE), investigator-initiated, study that will define the efficacy and safety of edoxaban compared with non-anticoagulant medical therapy (no antithrombotic therapy or antiplatelet monotherapy) for stroke/systemic embolism prevention in high-risk AF patients and previous intracranial hemorrhage. Intracranial hemorrhage includes intracerebral hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage and subdural hematoma. Recruitment will occur at 250-300 stroke research centres in North and South America, Europe and Asia over 24 months, where 1200 adult participants with high-risk AF (CHA2DS2-VASc score ≥2) and previous spontaneous or traumatic intracranial hemorrhage (while on or off antithrombotic therapy) will be randomly assigned to receive edoxaban 60/30 mg daily or to non-anticoagulant medical therapy (no antithrombotic therapy or antiplatelet monotherapy). Consenting participants will be followed to a common study end-date in this event-driven trial once 123 primary efficacy events (stroke) have accrued; anticipated to be about 12 months after the end of recruitment.

ENRICH-AF will assess the safety and efficacy of anticoagulant therapy in AF participants after intracranial hemorrhage, an area where there currently exists huge interest within the stroke and cardiology research communities. Demonstrating safety comparable with non-anticoagulant medical therapy in AF patients who are particularly at high risk for intracranial hemorrhage is likely to have a more far-reaching clinical impact than solely within the proposed study population. ENRICH-AF will be the "ultimate safety test" of anticoagulation of AF patients, providing reassuring evidence favoring more widespread use of anticoagulation for stroke prevention in AF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided
2. Age ≥45 years, at the time of signing the informed consent
3. Previous intracranial hemorrhage (symptomatic, spontaneous and non-traumatic non-lobar intraparenchymal or intraventricular hemorrhage, and symptomatic spontaneous or non-penetrating traumatic subdural hemorrhages) on or off antithrombotic therapy
4. Documented atrial fibrillation (paroxysmal, persistent, permanent)
5. CHA2DS2-VASc score ≥2

Exclusion Criteria:

1. Recent intracranial hemorrhage (within 14 days)
2. Secondary macrovascular, neoplastic or infectious causes of intracranial hemorrhage (except for antithrombotic treatment or non-penetrating traumatic subdural hemorrhages)
3. Isolated subarachnoid hemorrhage (convexity or basal); subarachnoid blood tracking onto convexity secondary to an intraventricular hemorrhage or as part of a multicompartment bleed in cases of traumatic subdural hemorrhages are eligible
4. Need for ongoing oral anticoagulant therapy for indication other than AF (e.g. mechanical heart valve, venous thromboembolic disease)
5. Need for ongoing antiplatelet therapy for indication where edoxaban would not be a suitable substitute
6. Plans for left atrial appendage occlusion
7. Estimated creatinine clearance (CrCl) < 15 mL/min
8. Platelet count less than 100,000mm3 at enrollment or other bleeding diathesis
9. Persistent, uncontrolled hypertension (systolic BP averaging >150 mmHg)
10. Chronic use of NSAID
11. Clinically significant active bleeding, including gastrointestinal bleeding
12. Lesions or conditions at increased risk of clinically significant bleeding, e.g. active peptic ulcer disease with recent bleeding, patients with spontaneous or acquired impairment of hemostasis
13. Antiphospholipid antibody syndrome
14. Hepatic disease associated with coagulopathy and clinically relevant bleeding risk
15. Known hypersensitivity to edoxaban
16. Estimated inability to adhere to study procedures
17. Pregnancy or breastfeeding
18. Estimated life expectancy < 6 months at the time of enrollment
19. Close affiliation with the investigational site; e.g. a close relative for the investigator, dependent person (e.g., employee or student of the investigational site)
20. Lobar intraparenchymal hemorrhage

    * Post menopausal female subjects must be amenorrheic for ≥12 months prior to screening or ≥6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) prior to screening. Women of childbearing potential must have negative serum pregnancy test within 7 days prior to randomization or urine pregnancy testing within 24 hours of randomization. Heterosexually active women of childbearing potential must use highly effective methods of contraception for 32 days after discontinuation (duration of study drug plus 30 days duration of one ovulatory cycle).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 948 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Stroke or Systemic Embolism | From randomization until the common study end date (average of 3 years)
  Stroke (composite of ischemic, hemorrhagic and unspecified) or systemic embolism
Major hemorrhage | From randomization until the common study end date (median 2 years)
  as defined byt the International Society on Thrombosis and Haemostasis (ISTH) criteria

SECONDARY OUTCOMES:
Ischemic stroke | From randomization until the common study end date (median 2 years)
  development of an acute neurologic deficit in conjunction with brain imaging consistent with acute/subacute ischemic stroke.
Cardiovascular death | From randomization until the common study end date (median 2 years)
  Death related to cardiovascular cause
Hemorrhagic stroke | From randomization until the common study end date (median 2 years)
  development of an acute neurologic deficit in conjunction with brain imaging consistent with acute/subacute intraparenchymal, intraventricular or subarachnoid hemorrhage
Disabling/fatal stroke | From randomization until the common study end date (median 2 years)
  Disabling stroke is defined as stroke resulting in a clinical outcome that is associated with a modified Rankin scale of 4 or 5. Fatal stroke is defined as death occurring within 30 days of stroke.
Composite of all stroke, myocardial infarction, systemic thromboembolism, or all-cause death | From randomization until the common study end date (median 2 years)
  Components of composite outcome (adjudicated) includes stroke (ischemic, hemorrhagic, and undefined stroke, TIA with positive neuroimaging),myocardial infarction, systemic thromboembolism or all-cause death. Incidence rate estimated as number of participants with incident events divided by cumulative at-risk time, where participant is no longer at risk once an incident event occurred
Net clinical benefit (composite of stroke, myocardial infarction, cardiovascular death, fatal bleeding, and symptomatic bleeding into a critical organ or area) | From randomization until the common study end date (median 2 years)
  Net clinical benefit is a composite of stroke, myocardial infarction, cardiovascular death, fatal bleeding, and symptomatic bleeding into a critical organ or area
modified Rankin Scale | 12 months
  mRS as measured at 12 month visit
All intracranial hemorrhage (intracerebral hemorrhage, intraventricular hemorrhage, subdural hematoma, subarachnoid hemorrhage) | From randomization until the common study end date (median 2 years)
  Intracranial hemorrhage as defined by Signs or symptoms associated with an epidural, subdural, subarachnoid, intraparenchymal or intraventricular hemorrhage on computed tomography (CT) or MRI scan, or as demonstrated by surgery or autopsy.
Fatal intracranial hemorrhage | From randomization until the common study end date (median 2 years)
  Inctracranial hemorrhage defined as Signs or symptoms associated with an epidural, subdural, subarachnoid, intraparenchymal or intraventricular hemorrhage on computed tomography (CT) or MRI scan, or as demonstrated by surgery or autopsy with death occurring within 30 days of stroke
Subdural hemorrhage | From randomization until the common study end date (median 2 years)
  Subdural hemorrhage as defined as Signs or symptoms associated with a subdural hemorrhage on computed tomography (CT) or MRI scan, or as demonstrated by surgery or autopsy
Hospitalization for any cause | From randomization until the common study end date (median 2 years)
  Minimum of one overnight stay in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Shoamanesh, MD, FRCPC, Principal Investigator — Population Health Research Institute
Locations (152):
- United States (10):
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Presence Care Transformation Corporation, Lisle, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - New York Presbyterian - Queens, Queens, New York
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The University of Texas at Austin, Dell Medical School, Austin, Texas
  - Texas Tech University Health Sciences Center at El Paso, El Paso, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Argentina (5):
  - Stat Research S.A., Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (FLENI), Buenos Aires
  - Hospital Policial Churruca-Visca, Buenos Aires
  - Centro Instituto Neurologico Salta, Salta
- Austria (4):
  - Medical University of Innsbruck, Innsbruck
  - Institut für Akutneurologie und Stroke Unit (IANS), Landeskrankenhaus Feldkirch, Rankweil
  - Medical University of Vienna, Dept. of Neurology, Vienna
  - Salzkammergutklinikum Vöcklabruck, Vöcklabruck
- Belgium (10):
  - Erasme Hospital, Brussels
  - UZ Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Hospital, Hasselt
  - Groeninge Hospital, Kortrijk
  - UZ Leuven, Leuven
  - Clinique CHC MontLégia, Liège
  - AZ Damiaan, Ostend
  - AZ Delta, Roeselare
- Canada (18):
  - Brandon Regional Health Centre, Brandon
  - University of Calgary / Foothills Medical Centre, Calgary
  - Centre Intégré Universitaire de Santé et de Services Sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi
  - University of Alberta Hospital, Edmonton
  - Nova Scotia Health Authority, Halifax
  - Hamilton Health Sciences, Hamilton
  - Kingston General Hospital, Kingston
  - London Health Science Centre - University Hospital, London
  - CHUM Centre Hospitalier de l'Université de Montréal, Montreal
  - McGill University Health Centre, Montreal
  - The Ottawa Hospital Research Institute, Ottawa
  - The Rhema Research Institute, Owen Sound
  - CHUL Pavillon Enfant-Jésus, Québec
  - University of Saskatchewan, Saskatoon
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay
  - Sunnybrook Health Science Centre, Toronto
  - University Health Network - Toronto Western Hospital, Toronto
  - Canadian Cardiac Research Centre, Windsor
- China (8):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Punan Hospital, Shanghai
  - Shanghai Blue Cross Brain Hospital, Shanghai
  - Shanghai East Hospital, Tongji University, Shanghai
  - Shanghai Fengcheng Hospital, Shanghai
  - Xinhua Hospital, Chongming Branch, Shanghai
  - Yangpu Hospital, Tongji University, Shanghai
  - The First People's Hospital of Shenyang, Shenyang
- Czechia (3):
  - St. Anne's University Hospital, Brno
  - Neurological Department, General Hospital of Jihlava, Jihlava
  - Cerebrovaskularni poradna s.r.o., Ostrava
- Egypt (8):
  - Fayoum General Hospital, Al Fayyum
  - Mansoura University Hospital, Al Mansurah
  - Alexandria University Hospital, Alexandria
  - Beni Suef University Hospital, Banī Suwayf
  - Ain Shams Specialized Hospital, Cairo
  - Ain Shams University Hospital, Cairo
  - Tanta University Hospital, Tanta
  - Zagazig University Hospital, Zagazig
- Germany (14):
  - Charité - University Medicine Berlin, Berlin
  - Dresden University Hospital "Carl Gustav Carus", Dresden
  - Universitätsklinikum Essen, Essen
  - Klinikum Friedrichshafen, Friedrichshafen
  - University Medicine Goettingen, Goettigen
  - Martha-Maria Hospital, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum Main-Spessart, Krankenhaus Lohr, Lohr
  - Klinik fur Neurologie, UKSH campus Lubeck, Lübeck
  - Medical Faculty Mannheim, Heidelberg University, Mannheim
  - Westfalische Wilhelms-Universitat Munster, Münster
  - Klinikum Osnabrück; Neurologie, Osnabrück
  - Department of Neurology, Klinikum Vest, Recklinghausen
  - Universitätsklinikum Tübingen, Tübingen
- India (17):
  - Zydus Hospitals & Healthcare Research Pvt. Ltd., Ahmedabad
  - Shree Krishna Hospital and Pramukhswami Medical College, Anand
  - Bangalore Baptist Hospital, Bangalore
  - Fortis Hospital Ltd, Bangalore
  - Mazumdar Shaw Medical Center - Unit of Narayana Health, Bangalore
  - St. John's Medical College Hospital, Bangalore
  - Post Graduate Institute of Medical Education &Research, Chandigarh
  - Sikkim Manipal Institute of Medical Sciences, Gangtok
  - GNRC Hospitals, Guwahati
  - Bangur Institute of Neurosciences, Kolkata
  - Caritas Hospital, Kottayam
  - Christian Medical College & Hospital, Ludhiāna
  - Dhadiwal Hospital in coalition with Shreeji Healthcare, Nashik
  - Bharati Vidyapeeth (DTU) Medical College & Hospital, Pune
  - Nanjappa Hospital, Shimoga
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Thiruvananthapuram
  - Rhythm Heart Institute, Vadodara
- Nepal (9):
  - Chitwan Everest Asptalal Private limited, Bharatpur
  - Chitwan Medical College Teaching Hospital, Bharatpur
  - Nobel Medical College & Teaching Hospital, Biratnagar
  - B P Koirala Institute of Health Sciences, Dharān
  - B & C Medical College Teaching Hospital & Research Centre Pvt. Ltd., Jhapa
  - Annapurna Neurological institute and allied sciences, Kathmandu
  - Grande International Hospital, Kathmandu
  - Kathmandu Medical College, Kathmandu
  - Upendra Devkota Memorial-National Institute of Neurological and Allied Sciences (UDMNINAS), Kathmandu
- CHULN-Hospital Santa Maria, Lisbon, Portugal
- Spain (16):
  - Coruña University Hospital, A Coruña
  - University Hospital of Albacete, Albacete
  - Instituto de Investigacion Sanitaria Biocruces, Barakaldo
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu Isant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario de Cáceres, Cáceres
  - Hospital Donostia - Osidonostialdea, Donostia / San Sebastian
  - Hospital u Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramón y Cajal, Madrid
  - La Paz Univerity Hospital, Madrid
  - Hospital Universitario Central de Asturias-Finba, Oviedo
  - Hospital Universitario son Espases, Palma de Mallorca
  - Hospital Universitari i Politécnic La Fe., Valencia
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital, University Hospital Bern, Bern
- United Kingdom (27):
  - Aberdeen Royal Infirmary, NHS Grampian, Aberdeen
  - Nevill Hall Hospital, Abergavenny
  - NHS Lanarkshire Health Board - Monklands Hospital, Airdrie
  - Arrowe Park Hospital, Birkenhead
  - The Royal Bournemouth Hospital, Bournemouth
  - Bradford Teaching Hospitals NHS Foundation Trust, at Bradford Royal Infirmary, Bradford
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospital of Wales, Cardiff
  - East Suffolk and North Essex NHS Foundation Trust, at Colchester Hospital, Colchester
  - Edinburgh Royal Infirmary, Edinburgh
  - Queen Elizabeth Hospital - Gateshead Health NHS Foundation Trust, Gateshead
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - LNWUH - Northwick Park Hospital, Harrow
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - Victoria Hospital Kirkcaldy, Kirkcaldy
  - Homerton University Hospital, London
  - King's Mill Hospital, Mansfield
  - The South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Morriston Hospital, Morriston
  - Royal Preston Hospital, Preston
  - Royal Berkshire NHS Foundation Trust, Reading
  - Royal Cornwall Hospital, Truro
  - Hillingdon Hospital, Uxbridge
  - Southend University Hospital Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea
  - Yeovil District Hospital, Yeovil

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170